CLINICAL TRIAL: NCT02625584
Title: Reading Together: How to Promote Children's Language Development Using Family-based Shared Book Reading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caroline Rowland (Other)
Responsible Party: Sponsor-Investigator, Caroline Rowland, Professor, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RETH000849
Record Dates: First submitted 2015-11-24; First posted 2015-12-09 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Language Development
Keywords: Shared Book Reading; Dialogic Reading; Language Development; Syntax; Vocabulary; Young Children; Randomised Control Trial; Language Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shared Reading Control (Other): Reading Together - Shared Reading Control. The intervention will run for six weeks and the caregivers will be provided with books to read with their children. Caregivers will not be trained to read with their child. The caregivers will be asked to read two books to their child five times a week. Caregivers will keep a reading diary and audio record all shared book reading sessions with their child.
  Interventions: Behavioral: Reading Together - Shared Reading Control
- Dialogic Reading (Experimental): Reading Together - Dialogic Reading. The intervention will run for six weeks and the caregivers will be provided with books to read with their children. Caregivers will be trained to read with their child using a dialogic reading style. The caregivers will be asked to read two books to their child five times a week. Caregivers will keep a reading diary and audio record all shared book reading sessions with their child.
  Interventions: Behavioral: Reading Together - Dialogic Reading
- Pausing for Reading (Experimental): Reading Together - Pausing for Reading. The intervention will run for six weeks and the caregivers will be provided with books to read with their children. Caregivers will be trained to read with their child using a style which involves pausing, recasting and open questioning. The caregivers will be asked to read two books to their child five times a week. Caregivers will keep a reading diary and audio record all shared book reading sessions with their child.
  Interventions: Behavioral: Reading Together - Pausing for Reading

INTERVENTIONS:
Behavioral: Reading Together - Pausing for Reading
  Arms: Pausing for Reading
Behavioral: Reading Together - Dialogic Reading
  Arms: Dialogic Reading
Behavioral: Reading Together - Shared Reading Control
  Arms: Shared Reading Control

SUMMARY:
The aim of this project is to determine how shared reading promotes child language development, and to use this knowledge to make it an effective language-boosting tool for children from all social and economic backgrounds.

DETAILED DESCRIPTION:
Two interventions will be created which are intended to boost children's vocabulary and grammar abilities, and will be assessed on how they are implemented by caregivers across different socio economic groups, and how they affect children's development of these language skills. Previous research has found dialogic reading interventions to be less effective for children from low socio-economic backgrounds. This project will investigate whether a shared reading intervention, designed to require less of a behaviour change from caregivers than dialogic reading, can be used to effectively boost vocabulary and grammar development in children across the whole socio-economic spectrum.

ELIGIBILITY:
Inclusion Criteria:

* All families will be included unless they fit the exclusion criteria.

Exclusion Criteria:

* Children born before 37 weeks gestation (premature)
* Children who weighed less than 5lb 9oz at birth (low birth weight)
* Children who have had an ear infection/glue ear for longer than 3 months, 4-6 ear infections within a 6 month period or another identified hearing problem (e.g. at newborn hearing screening)
* Children with an identified developmental disability (e.g. Cerebral Palsy, Autism Spectrum Disorder, Fragile X syndrome, Muscular dystrophy, Di George syndrome, Down's syndrome, Williams syndrome)
* Children with a hearing or visual impairment
* Children who hear another language (not English) for 1 day or more in a typical week (please note that this also excludes children of parents who do not speak English)
* Children whose parents have a learning disability which puts their children at risk of language delay and excludes the parents from giving informed consent on their own and on their children's behalf.

Ages: 30 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in baseline language skills (PLS-5) | Baseline and 6 weeks
  The Preschool Language Scale Fifth Edition (PLS-5) Will be administered. This is a published standardized measure of the language knowledge of individual children. The investigators will use both the Auditory Comprehension and Expressive Communication scales to measure vocabulary and grammar knowledge. The PLS-5 standard scores are based on a mean of 100 with a standard deviation of 15. Scores between 85 and 115 are considered to be within the normal range.

SECONDARY OUTCOMES:
Change in baseline syntax comprehension (CELF Preschool-2 UK) | Baseline and 6 weeks
  The Clinical Evaluation of Language Fundamentals - Preschool 2 UK (CELF Preschool-2) will be administered. This is a published standardized measure of the language knowledge of individual children. The investigators will use the 'Sentence Structure' subtest. This will allow measurement of the children's understanding of a range of simple and complex sentence structures. A sentence is read to the child and the child chooses, from a set of pictures, which picture ''goes with'' that sentence.
Change in baseline caregiver dialogic reading behaviour | Baseline and 6 weeks
  10 minute video recordings of the dyads reading books at baseline and 6 weeks will be analysed for the number of target dialogic reading behaviours. This will allow measurement of the caregiver's dialogic reading behaviour pre- and post-intervention.
Change in baseline caregiver pause reading behaviour | Baseline and 6 weeks
  10 minute video recordings of the dyads reading books at baseline and 6 weeks will be analysed for the number of target pause reading behaviours. This will allow measurement of the caregiver's pause reading behaviour pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline F Rowland, PhD, Principal Investigator — The University of Liverpool
Locations (1):
- Liverpool Language Lab at the University of Liverpool, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Background] Manz PH , Hughes C , Barnabas E , Bracaliello C , Ginsburg-Block M. A descriptive review and meta-analysis of family-based emergent literacy interventions: To what extent is the research applicable to low-income, ethnic-minority or linguistically-diverse young children? Early Childhood Research Quarterly 25(4): 409-431, 2010.